CLINICAL TRIAL: NCT06723886
Title: Assessment of the Potential Antidiabetic Effects of Olive Pomace Oil in Diabetic or Prediabetic Subjects: Postprandial Study and Chronic Intervention
Brief Title: Antidiabetic Effect of Olive Pomace Oil
Acronym: OPODIABE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciencia y Tecnología de Alimentos y Nutrición (Other Government)
Collaborators: ICTAN-CSIC - Madrid - Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20232949; 253405 (Other: CSIC)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes Mellitus; Prediabetes (Insulin Resistance, Impaired Glucose Tolerance); Prediabetic State; Diabetes; Diabetes Mellitus
Keywords: Olive pomace oil; Diabetes; Prediabetes; Antidiabetic effect; Postprandial study; Chronic intervention; High-oleic acid sunflower oil
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Insulin Resistance; Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Crossover, controlled, randomized, blind study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olive pomace oil (Experimental): Consumption of olive pomace oil as the only dietary fat.
  Interventions: Dietary Supplement: Experimental arm: Olive pomace oil
- High-sunflower olive oil (Active Comparator): Consumption of high-oleic acid sunflower oil as the only dietary fat.
  Interventions: Dietary Supplement: High-oleic acid sunflower oil

INTERVENTIONS:
Dietary Supplement: Experimental arm: Olive pomace oil — Participants will consume during 8 weeks either the test oil (olive pomace oil) as the only dietary fat. They will consume 45 g/day of oil, using it in salads, fried foods, as spread on toasts, etc.
  Arms: Olive pomace oil
Dietary Supplement: High-oleic acid sunflower oil — Participants will consume during 8 weeks either the test active comparator oil (high-oleic acid sunflower oil) as the only dietary fat. They will consume 45 g/day of oil, using it in salads, fried foods, as spread on toasts, etc.
  Arms: High-sunflower olive oil

SUMMARY:
This clinical trial aims at assessing whether consumption of olive pomace oil in the diet may benefit persons with type 2 diabetes mellitus or persons at risk of developing the disease (prediabetic persons).

The main questions the study aims to answer are:

* May olive pomace oil prevent a high increase of blood glucose levels when consumed in a meal together with carbohydrates in diabetic/prediabetic patients?
* May olive pomace oil decrease fasting blood glucose levels of diabetic/prediabetic patients after consuming it daily?
* May daily consumption of olive pomace oil improve glucose homeostasis and other alterations like elevated blood lipids or inflammation, which also affect persons with diabetes or prediabetes?

Researchers will compare the effect of consuming olive pomace oil to the effects of a comparison oil (high-oleic acid sunflower oil).

Participants will:

In different days, they will consume white bread alone or the oils (olive pomace oil, high-oleic acid sunflower oil or extra virgin olive oil) spread on white bread and blood will be collected at different times during 2 h. This study to observe the increase of blood glucose after a carbohydrate-rich breakfast will be part of the so-called "postprandial" study, and will be conducted during 3 weeks, during which participants will consume corn oil on a daily basis.

Participants will also take part in the "chronic" study, that will last 22 weeks in total. During this study, they will firstly "wash" the effects of the oil they normally consume in their diets by consuming corn oil during 3 weeks. It is during these weeks when they will attend the Human Nutrition Unit (HNU) of ICTAN to carry on the "postprandial" study described in the previous paragraph.

After the initial 3 weeks, participants will consume olive pomace oil as the only oil in their diets during 8 weeks, "wash" its effects again by consuming corn oil during 3 weeks and then change to consume the other oil (high-oleic acid sunflower oil) during 8 weeks.

During the chronic study, they will visit the clinic once every 4 weeks for checkups and tests. They will refrain from eating other oils or specific fat-rich foods. Participants will also attend our phone calls to ask them what they ate the day before on different weeks during the study, and wear an accelerometer during 1 week to record their physical activity. They will keep a diary of the doses of insulin/metformin used and the blood glucose levels they measured at home.

DETAILED DESCRIPTION:
This trial comprises 2 studies in parallel, a postprandial study and a chronic intervention.

In the postprandial study, participants will attend the Human Nutrition Unit (HNU) of ICTAN in different days. During these visits, they will consume white bread (50 g) alone or with 10 g of extra virgin olive oil (EVOO), olive pomace oil (OPO) or high-oleic acid sunflower oil (HOSO). A nurse will insert a catheter in the non-prevailing arm and collect fasting blood (0 h) and blood samples 1 and 2 h after consuming the bread/oil to measure the postprandial glycemic/insulinemic response, as well as incretins (GLP-1, GIP). Blood lipids will also be determined. These visits will be carried out during the 3-week run-in period prior to the chronic intervention, when the EVOO and control (white bread) tests will be carried out (weeks 1 and 2, respectively). Then, coinciding with the first day of the chronic intervention, participants will consume either OPO or HOSO as corresponding to the randomized allocation to each oil. The other postprandial test will be carried out at the beginning of the second intervention after crossover and wash-out, thus avoiding additional visits and discomfort to the participants.

The chronic study is a crossover, randomized, blind, clinical trial. After a 3-week run-in during which participants will consume corn oil as the only dietary oil, they will be randomly allocated to one of each intervention arms, OPO or HOSO, each lasting 8 weeks. Then, a 3-week wash-out period with corn oil will follow before changing to consuming the other oil.

During the study, participants should avoid other oils and fats such as olives, sunflower seeds, butter, margarine, nuts or avocados.

During the chronic intervention, participants will visit the HNU at the beginning (week 1), middle (week 4) and at the end (week 8) of each intervention arm. A nurse will collect a fasting blood sample and measure blood pressure. An analysis of body weight and body composition (anthropometric and bioimpedance measurements) will be performed. Participants should maintain their habitual diet and exercise level throughout the study; diet will be monitored by periodic 24-h recall questionnaires (a trained member of the team will phone participants on 3 different days (including a festive one) before each visit to the HNU to enquire what they ate the previous day). In addition, a physical activity questionnaire will be completed at the beginning of the study and, on each intervention arm, participants will carry during 7 days an accelerometer to monitor real physical activity.

Biochemical, hormonal and inflammatory markers will be measured in blood samples to assess the potential effect of olive pomace oil on different outcomes of relevance in the management of blood glucose in diabetic/prediabetic persons, including glucose homeostasis, insulin resistance, blood lipid levels, liver function, different hormones, incretins, adipokines, pro- and anti-inflammatory cytokines, on integrity of the intestinal barrier.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose between 100-126 mg/dL and/or
* Glycated haemoglobin (HbA1c) between 5.7-6.4% and/or
* Diabetic persons with Fasting blood glucose >126 mg/dL and/or
* Diabetic persons with Glycated haemoglobin (HbA1c) > 6.4%

Exclusion Criteria:

* Kidney or liver diseases
* Gastrointestinal diseases (irritable bowel syndrome, Crohn disease, chronic bowel inflammation)
* Food allergies/intolerances
* Vegetarians/vegans
* Smoking
* Pregnant or lactating women
* On prescription drugs other than for hypertension/thyroid/dyslipidemia/glucose control, or changes in dosage in the last 3 months
* Consumption of vitamins, dietary supplements or nutraceuticals

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | From enrollment to the end of each treatment at 8 weeks
  Change of fasting blood glucose levels at the end of the chronic intervention
Postprandial blood glucose response | From enrollment until week 14 of the study
  Change of postprandial blood glucose levels after consuming white bread with oil in comparison with white bread only.
  Blood will be collected at 0 h and 1 and 2 h after consuming the bread alone or with the corresponding oil. Olive pomace oil (active comparator) and high-oleic acid sunflower oil (active comparator) will be tested. Only in this postprandial study extra virgin olive oil will also be tested as a positive control (at the beginning of the run-in), along with white bread only (at week 2 of the run-in). Test/comparator oils will be assessed at the beginning of each arm, week 1 of each intervention arm (corresponding to weeks 4 and 14 of the study).

SECONDARY OUTCOMES:
Insulin levels | From enrollment to the end of each treatment at 8 weeks
  Change in fasting blood insulin levels at the end of the chronic intervention
Insulin resistance | From enrollment to the end of each treatment at 8 weeks
  Change in homeostasis model assessment (HOMA) of insulin resistance (HOMA-IR) at the end of the chronic intervention
Insulin sensitivity | From enrollment to the end of each treatment at 8 weeks
  Change in quantitative insulin levels sensitivity check index (QUICKI) at the end of the chronic intervention. Higher score in QUICKI means a better outcome compared to initial values.
Glycated hemoglobin | From enrollment to the end of each treatment at 8 weeks
  Change in blood levels of glycated hemoglobin (HbA1c) at the end of the chronic intervention
Beta-cell function | From enrollment to the end of each treatment at 8 weeks
  Change in homeostasis model assessment (HOMA) of beta-cell function (HOMA-B) at the end of the chronic intervention
Postprandial insulin response | From enrollment to week 14 of the study
  Change of postprandial blood insulin levels after consuming white bread with oil in comparison with white bread only.
  Blood will be collected at 0 h and 1 and 2 h after consuming the bread alone or with the corresponding oil. Olive pomace oil (active comparator) and high-oleic acid sunflower oil (active comparator) will be tested. Only in this postprandial study extra virgin olive oil will also be tested as a positive control (at the beginning of the run-in), along with white bread only (at week 2 of the run-in). Test/comparator oils will be assessed at the beginning of each arm, week 1 of each intervention arm (corresponding to weeks 4 and 14 of the study).
Postprandial incretins | From enrollment to week 14 of the study
  Change of postprandial levels of GLP-1 and GIP after consuming white bread with oil in comparison with white bread only.
  Blood will be collected at 0 h and 1 and 2 h after consuming the bread alone or with the corresponding oil. Olive pomace oil (active comparator) and high-oleic acid sunflower oil (active comparator) will be tested. Only in this postprandial study extra virgin olive oil will also be tested as a positive control (at the beginning of the run-in), along with white bread only (at week 2 of the run-in). Test/comparator oils will be assessed at the beginning of each arm, week 1 of each intervention arm (corresponding to weeks 4 and 14 of the study).
Postprandial blood lipids | From enrollment to week 14 of the study
  Change of postprandial blood lipid levels after consuming white bread with oil in comparison with white bread only.
  Blood will be collected at 0 h and 1 and 2 h after consuming the bread alone or with the corresponding oil. Olive pomace oil (active comparator) and high-oleic acid sunflower oil (active comparator) will be tested. Only in this postprandial study extra virgin olive oil will also be tested as a positive control (at the beginning of the run-in), along with white bread only (at week 2 of the run-in). Test/comparator oils will be assessed at the beginning of each arm, week 1 of each intervention arm (corresponding to weeks 4 and 14 of the study).

OTHER OUTCOMES:
Blood lipids | From enrollment to the end of each treatment at 8 weeks
  Change in serum levels of total cholesterol or LDL-cholesterol or HDL-cholesterol or triglycerides or apolipoprotein A1 or apolipoprotein B at the end of the chronic intervention
Inflammatory cytokines | From enrollment to the end of each treatment at 8 weeks
  Change in the levels of C-reactive protein (CRP), or pro-inflammatory cytokines (tumor necrosis factor-alpha (TNF-a), or interferon gamma (IFN-g), or interleukin (IL)-1beta (IL-1b), or IL-2, or IL-5, or IL-6, or IL-7, or IL-8, or IL-13)) or anti-inflammatory cytokines IL-4 or IL-10 at the end of the chronic intervention
Liver function | From enrollment to the end of each treatment at 8 weeks
  No changes in serum levels of alanine transferase (ALAT), or aspartate transferase (ASAT) or gamma-glutamyl transferase (GGT) at the end of the chronic intervention
Hormones, incretins and adipokines levels | From enrollment to the end of each treatment at 8 weeks
  Changes in serum levels of C peptide or glucagon or fibroblast growth factor 21 (FGF21) or glucagon inhibitory peptide (GIP) or glucagon-like peptide type 1 (GLP-1) or ghrelin or leptin or resistin or plasminogen activator inhibitor type 1 (PAI-1) or visfatin or adiponectin or adipsin or dipeptidyl peptidase IV (DPP IV) at the end of the chronic intervention
Intestinal barrier function | From enrollment to the end of each treatment at 8 weeks
  Changes in blood levels of lipopolysaccharide (LPS) or zonulin at the end of the chronic intervention

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bravo, Professor, Principal Investigator — ICTAN-CSIC
Locations (1):
- Institute of Food Science, Technology and Nutrition (ICTAN-CSIC), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Interesting researchers may contact the principal investigator
Supporting Information: Study Protocol, ICF
Time Frame: After completion of the study and publication of results
Access Criteria: Justified request to the principal investigator